CLINICAL TRIAL: NCT03869424
Title: Influence of Expectations on Rumination: An Experimental Investigation
Brief Title: Influence of Expectations on Rumination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-05k
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Expectations Group (Experimental): Participants receive a nasal spray that is in fact a placebo. However, they are told that it protects from rumination. They take the nasal spray once in the laboratory.
  Interventions: Other: Active Placebo labelled as antidepessant
- No-treatment control group (No Intervention): Participants do not receive the nasal spray.

INTERVENTIONS:
Other: Active Placebo labelled as antidepessant — Participants receive an active nasal spray that is in fact a placebo.
  Arms: Positive Expectations Group

SUMMARY:
The study tries to identify whether positive expectations, induced with an active placebo nasal-spray, have effects on rumination.

DETAILED DESCRIPTION:
Healthy volunteers are informed that a new application method for an antidepressant, specialised on protecting from rumination, would be tested. They will randomly be assigned to the treatment group (taking the antidepressant which is in fact an active placebo) or the no treatment control group (not taking a placebo). Then sad mood is induced by mood-suggestive music and negative autobiographic recall. Then participants in the experimental group take the "medication". Afterwards both groups are asked to focus on emotion-focused, symptom-focused and self-focused thoughts to induce rumination (e.g. "Think about what your feelings might mean."). Sadness will be assessed before and after the negative recall task and also after the rumination induction. State Rumination will be assessed before the recall task and after the rumination induction.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* fluent in German language

Exclusion Criteria:

* mental disorders
* allergic to capsaicin
* allergic to sesame oil
* intake of psychopharmacological drugs in the last four weeks
* intake of illegal drugs in the last two weeks
* consumption of alcohol in the last twelve hours
* students in medicine, pharmacy, or psychology
* completed studies in medicine, pharmacy or psychology
* current pregnancy or lactation
* cardio vascular disease
* kidney disease
* liver disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-08-14 (Actual)

PRIMARY OUTCOMES:
Change in State Rumination (Fragebogen zur Erfassung aktueller Ruminationsneigung) | At baseline and after the rumination induction. Each assessment is taking 5 Minutes, in total 10 minutes.
  German questionnaire of 10 Items, e.g.: "I get lost in ruminative thoughts.", "I am present in this situation.", "My thoughts are focused on the past.".All Items will be rated on a visual analogue scale from 0 (not at all) to 10 (very much).
Change in Positive and Negative Affect Schedule (PANAS-X) | At baseline, after the negative biographical recall and after the rumination induction, each assessment is taking 3 minutes, in total 9 minutes.
  Items of PANAS-X: Sadness Score ("sad", "blue", "downhearted", "alone", "lonely") and Items "Surprised", "concentrating", "happy". All Items will be rated on a visual analogue scale from 0 (not at all) to 10 (very much).

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Professor, Principal Investigator — Philipps-Univeristy of Marburg
Locations (1):
- Philipps-Universität Marburg, Marburg, Deutschland, Germany